CLINICAL TRIAL: NCT04646642
Title: Psychological Health, Coping Strategies and Preferences of David Grant USAF Medical Center COVID-19 Deployers: A Critical Needs Assessment
Brief Title: Psychological Health, Coping Strategies and Preferences of Military COVID-19 Deployers
Status: Completed | Type: Observational
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amanda Fox, Clinical Inquiry in Nursing Readiness Fellow, David Grant U.S. Air Force Medical Center
Other Study IDs: FWH20200203E
Record Dates: First submitted 2020-11-25; First posted 2020-11-30 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Coping Skills; Healthcare Workers; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposed research study aims to better understand COVID deployer needs. The study, informally referred to as Project COPE, asks David Grant U.S. Air Force Medical Center (DGMC) members who deployed in support of COVID-19 operations to complete a needs assessment questionnaire. The purpose of this study is to understand the stressful experiences of our COVID Theater Hospital (CTH) deployers, the typical coping strategies used and recommended preferences for support so that the investigators can provide the best evidence-based resources for post-deployment and to aid future CTH deployers.

DETAILED DESCRIPTION:
Objective: This study focuses on exploring David Grant USAF Medical deployer psychological status and the coping skills utilized during deployment as well as a needs assessment of preferred coping resources.

Specific Aims:

* Aim 1: Describe the post-deployment state of psychological health for COVID-19 Theater Hospital (CTH) deployers
* Aim 2: Identify the deployer identified COVID-19-related stressors reported post deployment
* Aim 3: Identify coping and cognition regulating strategies used by deployers in response to COVID-19 deployment stressors
* Aim 4: Identify deployer coping resource preferences for future deployment support packages

Methods: Recruitment of eligible participants will include email invitations, packets with pre-printed needs assessment folders placed next to posters, flyers, and briefing at DGMC events. Eligible participants (n=160) returning from COVID Theater Hospital (CTH) deployment (est. Oct 2020) will receive a needs assessment that includes:

1. Patient Health Questionnaire-2 (PHQ-2) is a 2-item screening tool for depression that uses the first two items from the 9-item Patient Health Questionnaire. Respondents are asked to report symptom frequency ranging from 0 (not at all) to 3 (nearly every day) for the following questions, "Over the last 2 weeks, how often have you been bothered by any of the following problems: 1) little interest or pleasure in doing things, and 2) feeling down, depressed, or hopeless?" Total scores exceeding 2 suggest a positive depression screening. Participants who screen positive should be evaluated with the PHQ-9 to identify diagnostic depressive disorder criteria. It is important to note that all CTH deployers will complete a PHQ-9 during their post-deployment health assessment. Construct and criterion validity were established in a sample of 6000 primary care and obstetrics patients where the PHQ-2 score had a sensitivity of ≥ 83% and a specificity of 92% for major depression. A PHQ-2 score of 3 was identified as the optimal cut point as indicated by likelihood ratio and receiver operator characteristic analysis (Kroenke, Spitzer, & Williams, 2003). This tool provides a brief, practical, valid, and reliable screening instrument.
2. Generalized Anxiety Disorder-2 (GAD-2) is a 2-item screening tool for Generalized Anxiety Disorder. The tool asks respondents to report symptom frequency ranging from 0 (not at all) to 3 (nearly every day) for the following two questions: "Over the last 2 weeks, how often have you been bothered by the following problems:1) Feeling nervous, anxious or on edge, and, 2) Not being able to stop or control worrying?" A total score of 3 points or greater identifies a positive screen and warrants further diagnostic evaluation with the GAD-7 for Generalized Anxiety Disorder criteria. It is important to note that all CTH deployers will complete a GAD-7 during their post-deployment health assessment. The GAD-2 was validated in a randomized sample of 965 primary care patients demonstrating a sensitivity of 86% and specificity of 83% with an 0.908 area under the curve (95% CI) for a diagnosis of Generalized Anxiety Disorder (Kroenke, Spitzer, Williams, Monahan, & Lö, 2007). This tool provides a brief, practical, valid, and reliable screening instrument.
3. Pittsburgh Sleep Quality Index-Addendum for PTSD (PSQI-A) is a 7-item questionnaire used to examine disruptive nocturnal behaviors (hot flashes, nervousness, traumatic memories, anxiety, bad dreams, terror/screaming, acting out dreams) common in adults with PTSD. Response items are endorsed for frequency (not during the past month, less than once a week, once or twice a week, three or more times a week). Good internal consistency and convergent validity were demonstrated with anxiety, depression, sleep quality, combat exposure, and PTSD symptoms. The PSQI-A had a Cronbach's #= 0.72 and an average inter-item correlation r = 0.44 (range 0.27-0.57) with the PSQI-A total score. Area under the curve was 0.81, for a cut point ≥ 4 resulting in 71% sensitivity, 82% specificity, and 60% positive and 83% negative predictive value for clinically diagnostic PTSD purposes and a 74% correct classification (Insana, Hall, Buysse, & Germain, 2013). Sleep disturbances reflect a core dysfunction underlying PTSD. The PSQI-A is a valid instrument for PTSD applicable to both clinical and research settings.It is important to note that all CTH deployers will complete a Post-Traumatic Stress Disorder screening during the post-deployment health assessment.
4. Deployer Identified COVID-19 Stressors. Currently there are no valid and reliable instruments specific to COVID-19 distress. Given this is a novel pandemic, investigators requested deployers to list top 3 stressors experienced during deployment. Participants rated listed items as: 1-no distress, 2-mildy distressing, 3-distressing 4-very distressing, and 5-extremely distressing.
5. The Brief Coping Orientation to Problems Experienced (Brief COPE) is a 28-item multidimensional measure of 14 strategies (humor, positive reframing, acceptance, active coping, planning, behavioral disengagement, self-distraction, substance use, denial, self-blame, venting, emotional support, instrumental support, religion) used for coping or regulating cognitions in response to stressors. This abbreviated inventory (based on the complete 60-item COPE Inventory) is comprised of items that assess the frequency with which a person uses different coping strategies rated on a scale from 0-"I haven't been doing this at all" to 4-"I've been doing this a lot." (Amoyal et al., 2011). Investigators eliminated two items that deal with drugs and alcohol to maintain the eligibility of exempt protocol status.
6. COVID-19 Coping Strategy and Resource Inventory is an 18-item resource inventory developed by the DGMC research team to assess preferred strategic resources to manage COVID-19-related stressors. The inventory includes 5 categories of coping resources: 1) interactive [exercise, spiritual, social, mental health visit], 2) self-help videos/webinars, 3) mobile applications, 4) electronic toolkits, 5) podcasts.
7. Demographic questionnaire includes 10 questions regarding individual deployer sex, COVID-19 risk status, mental health risk status, COVID-19 risk status of any family members at home, years of experience in current occupation and specific healthcare role, typical work setting at DGMC, any recent deployments

Study participation will occur through a single collection of anonymous self-report measures using paper pencil which will be completed with an anticipated time burden of under 15 minutes (based on preliminary practice trials) and returned to locked drop-boxes strategically placed on four inpatient/outpatient areas.

Results: Findings will inform the development of a DGMC COVID-19 healthcare worker psychological coping and well-being toolkit.

ELIGIBILITY:
Inclusion Criteria:

* The eligible participant group includes David Grant United States Air Force (USAF) Medical Center Active Duty personnel:

  1. Medical technicians (4N)
  2. Liaison officers (LNO's)
  3. Nurses
  4. Physician assistants
  5. Advanced practice nurses
  6. Respiratory therapists
  7. Psychologists
  8. Social workers
  9. Chaplains
  10. Physicians
* Deployed in July 2020, under the command of Col Justin Nast and the COVID Theater Hospital (CTH) in support of the following civilian facilities:

  1. Adventist Health Lodi Memorial Hospital, Lodi, CA
  2. Eisenhower Medical Center, Rancho Mirage, CA
  3. Community Regional Medical Center, Fresno, CA
  4. Kaweah Delta Health Care, Visalia, CA
  5. Adventist Health Dameron Hospital, Stockton, CA
  6. Adventist Health Hanford, Hanford, CA
  7. Los Angeles County-University of Southern California (LA County-USC) Medical Center, Los Angeles, CA
  8. Harbor-University of California Los Angeles (UCLA) Medical Center, Torrance, CA

Exclusion Criteria:

* Activated guard, reserve, or civilian healthcare deployers in support of COVID-19
* Active duty healthcare deployers from MTF's other than DGMC in support of California (CA) civilian hospitals other than the eight facilities named in the above inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Active duty healthcare workers assigned to David Grant U.S. Air Force Medical Center (DGMC) who deployed in July 2020, under the command of Col Justin Nast and the COVID Theater Hospital (CTH), in support of 8 civilian California hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Positive Patient Health Questionnaire-2 (PHQ-2) | 1-2 months
  Describe the frequencies of positive screen for depression based on total score >/= 3 on PHQ-2. The PHQ-2 is a 2-item screening tool for depression that uses first 2 items from PHQ-9. Scale 0 (not at all) to 3 (nearly every day), 0 is better and 3 worse. Total scores exceeding 2 suggest a positive depression screening. This tool provides a brief, practical, valid, and reliable screening instrument.
Positive PHQ-2 + High risk COVID physical condition | 1-2 months
  Describe the frequencies and percentages of positive screened PHQ-2 individuals who also responded YES for self-reported high-risk COVID physical conditions on demographic questionnaire. The PHQ-2 is a 2-item screening tool for depression that uses first 2 items from PHQ-9. Scale 0 (not at all) to 3 (nearly every day), 0 is better and 3 worse. Total scores exceeding 2 suggest a positive depression screening. This tool provides a brief, practical, valid, and reliable screening instrument. The demographic questionnaire consist of 10 questions, one is COVID-19 risk status. A YES response to "Do you have any underlying physical health conditions that place you in a high-risk COVID category would be included in this measure.
Positive PHQ-2 + pre-existing mental health conditions | 1-2 months
  Describe the frequencies and percentages of positive screened PHQ-2 individuals who also responded YES for self-reported pre-existing mental health conditions on demographic questionnaire. The PHQ-2 is a 2-item screening tool for depression that uses first 2 items from PHQ-9. Scale 0 (not at all) to 3 (nearly every day), 0 is better and 3 worse. Total scores exceeding 2 suggest a positive depression screening. This tool provides a brief, practical, valid, and reliable screening instrument. The demographic questionnaire consist of 10 questions, one is mental health risk status. A YES response to "Do you have any underlying mental health concerns (anxiety, depression, difficulty sleeping, etc.), or have you visited a mental health professional in the past 6 months?" would be included in this measure.
Positive Generalized Anxiety Disorder-2 (GAD-2) | 1-2 months
  Describe the frequencies of positive screen for depression based on total score >/= 3 on GAD-2. The GAD-2 is a 2-item screening tool for Generalized Anxiety Disorder. Scale 0 (not at all) to 3 (nearly every day), 0 is better and 3 worse. A total score of 3 points or greater identifies a positive screen and warrants further diagnostic evaluation with GAD-7 for Generalized Anxiety Disorder criteria. This tool provides a brief, practical, valid, and reliable screening instrument.
Positive GAD-2 + High risk COVID physical condition | 1-2 months
  Describe the frequencies and percentages of positive screened GAD-2 individuals who also responded YES for self-reported high-risk COVID physical conditions on demographic questionnaire. The GAD-2 is a 2-item screening tool for Generalized Anxiety Disorder. Scale 0 (not at all) to 3 (nearly every day), 0 is better and 3 worse. A total score of 3 points or greater identifies a positive screen and warrants further diagnostic evaluation with GAD-7 for Generalized Anxiety Disorder criteria. This tool provides a brief, practical, valid, and reliable screening instrument. The demographic questionnaire consist of 10 questions, one is COVID-19 risk status. A YES response to "Do you have any underlying physical health conditions that place you in a high-risk COVID category would be included in this measure.
Positive GAD-2 + pre-existing mental health conditions | 1-2 months
  Describe the frequencies and percentages of positive screened GAD-2 individuals who also responded YES for self-reported pre-existing mental health conditions on demographic questionnaire. The GAD-2 is a 2-item screening tool for Generalized Anxiety Disorder. Scale 0 (not at all) to 3 (nearly every day), 0 is better and 3 worse. A total score of 3 points or greater identifies a positive screen and warrants further diagnostic evaluation with GAD-7 for Generalized Anxiety Disorder criteria. This tool provides a brief, practical, valid, and reliable screening instrument. The demographic questionnaire consist of 10 questions, one is mental health risk status. A YES response to "Do you have any underlying mental health concerns (anxiety, depression, difficulty sleeping, etc.), or have you visited a mental health professional in the past 6 months?" would be included in this measure.
Positive Pittsburgh Sleep Quality Index-Addendum for PTSD (PSQI-A) | 1-2 months
  Describe the frequencies of positive screen for depression based on total score > 4 on PSQI-A. The PSQI-A is a 7-item questionnaire used to examine disruptive nocturnal behaviors common in adults with PTSD. Response items are endorsed for frequency. Scale 0 (not during the past month) to 4 (3 or more times a week), 0 is better and 4 worse. The PSQI-A is a valid instrument for PTSD applicable to both clinical and research settings.
Positive PSQI-A + High risk COVID physical condition | 1-2 months
  Describe the frequencies and percentages of positive screened PSQI-A individuals who also responded YES for self-reported high-risk COVID physical conditions on demographic questionnaire. The PSQI-A is a 7-item questionnaire used to examine disruptive nocturnal behaviors common in adults with PTSD. Response items are endorsed for frequency. Scale 0 (not during the past month) to 4 (3 or more times a week), 0 is better and 4 worse. The PSQI-A is a valid instrument for PTSD applicable to both clinical and research settings. The demographic questionnaire consist of 10 questions, one is COVID-19 risk status. A YES response to "Do you have any underlying physical health conditions that place you in a high-risk COVID category would be included in this measure.
Positive PSQI-A + pre-existing mental health conditions | 1-2 months
  Describe the frequencies and percentages of positive screened PSQI-A individuals who also responded YES for self-reported pre-existing mental health conditions on demographic questionnaire. The PSQI-A is a 7-item questionnaire used to examine disruptive nocturnal behaviors common in adults with PTSD by frequency. Scale 0 (not during the past month) to 4 (3 or more times a week), 0 is better and 4 worse. The demographic questionnaire consist of 10 questions, one is mental health risk status. A YES response to "Do you have any underlying mental health concerns (anxiety, depression, difficulty sleeping, etc.), or have you visited a mental health professional in the past 6 months?" would be included in this measure.
Deployer Identified COVID-19 Stressors | 1-2 months
  Describe the severity of deployer identified COVID-19 stressors. A tool that requests deployers to list top 3 stressors experienced during deployment. Participants rated listed items as: 1-no distress, 2-mildly distressing, 3-distressing, 4- very distressing, and 5-extremely distressing. Scale 0 (no distress) to 5 (extremely distressing), 0 is better and 5 worse.
Positive Brief Coping Orientation to Problems Experienced (Brief COPE) | 1-2 months
  Describe the prevalence of positive coping strategies by percentage based on scores >/= 3 (3-I've been doing this medium amount; 4-I've been doing this a lot) for items targeting: humor, positive reframing, acceptance, active coping, planning, emotional support, instrumental support, religion. The Brief COPE is a 28-item multidimensional measure of 14 strategies (those above, as well as, behavioral disengagement, self-distraction, substance use, denial, self-blame, venting) used for coping or regulating cognitions in response to stressors. This abbreviated inventory (based on the complete 60-item COPE Inventory) is comprised of items that assess the frequency with which a person uses different coping strategies rated on a scale from 0-"I haven't been doing this at all" to 4-"I've been doing this a lot." (Amoyal et al., 2011). 4 is better and 0 worse. Two items related to drugs and alcohol were eliminated to maintain the eligibility of exempt protocol status
Negative Brief Coping Orientation to Problems Experienced (Brief COPE) | 1-2 months
  Describe the prevalence of negative coping strategies by percentage based on scores >/= 3 (3-I've been doing this medium amount; 4-I've been doing this a lot) for items targeting: behavioral disengagement, self-distraction, substance use, denial, self-blame, venting. The Brief COPE is a 28-item multidimensional measure of 14 strategies (those above, as well as, humor, positive reframing, acceptance, active coping, planning, emotional support, instrumental support, religion) used for coping or regulating cognitions in response to stressors. This abbreviated inventory (based on the complete 60-item COPE Inventory) is comprised of items that assess the frequency with which a person uses different coping strategies rated on a scale from 0-"I haven't been doing this at all" to 4-"I've been doing this a lot." (Amoyal et al., 2011). 0 is better and 4 worse. Two items related to drugs and alcohol were eliminated to maintain the eligibility of exempt protocol status
COVID-19 Coping Strategy and Resource Inventory | 1-2 months
  Describe the frequency of preferred coping resources using the COVID-19 Coping Strategy and Resource Inventory. This is an 18-item resource inventory developed by our DGMC research team to assess preferred strategic resources to manage COVID-19-related stressors. The inventory includes 5 categories of coping resources: 1) interactive [exercise, spiritual, social, mental health visit], 2) self-help videos/webinars, 3) mobile applications, 4) electronic toolkits, 5) podcasts
Demographic questionnaire | 1-2 months
  Describe the demographic characteristics of the respondents using the demographic questionnaire. These are 10 questions regarding individual deployer sex, COVID-19 risk status, mental health risk status, COVID-19 risk status of any family members at home, years of experience in current occupation and specific healthcare role, typical work setting at DGMC, any recent deployments.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda A Fox, MSN, Principal Investigator — David Grant Medical Center, Travis Air Force Base; Laurie A Migliore, PhD, Principal Investigator — David Grant Medical Center, Travis Air Force Base
Locations (1):
- David Grant Medical Center (DGMC), Travis Air Force Base, California, United States

REFERENCES:
- [Background] Amoyal NR, Mason ST, Gould NF, Corry N, Mahfouz S, Barkey A, Fauerbach JA. Measuring coping behavior in patients with major burn injuries: a psychometric evaluation of the BCOPE. J Burn Care Res. 2011 May-Jun;32(3):392-8. doi: 10.1097/BCR.0b013e318217f97a. PMID 21562462
- [Background] Braquehais MD, Vargas-Caceres S, Gomez-Duran E, Nieva G, Valero S, Casas M, Bruguera E. The impact of the COVID-19 pandemic on the mental health of healthcare professionals. QJM. 2020 Jun 22:hcaa207. doi: 10.1093/qjmed/hcaa207. Online ahead of print. PMID 32569374
- [Background] Cacioppo JT, Reis HT, Zautra AJ. Social resilience: the value of social fitness with an application to the military. Am Psychol. 2011 Jan;66(1):43-51. doi: 10.1037/a0021419. PMID 21219047
- [Background] Cullen W, Gulati G, Kelly BD. Mental health in the COVID-19 pandemic. QJM. 2020 May 1;113(5):311-312. doi: 10.1093/qjmed/hcaa110. No abstract available. PMID 32227218
- [Background] The Depressed Project: Living Systematic Review of Mental Health in COVID-19 Retrieved August 27, 2020, https://www.depressd.ca/covid-19-mental-health
- [Background] Folkman S. Personal control and stress and coping processes: a theoretical analysis. J Pers Soc Psychol. 1984 Apr;46(4):839-52. doi: 10.1037//0022-3514.46.4.839. PMID 6737195
- [Background] Greenberg N. Mental health of health-care workers in the COVID-19 era. Nat Rev Nephrol. 2020 Aug;16(8):425-426. doi: 10.1038/s41581-020-0314-5. PMID 32561871
- [Background] Hawkley LC, Thisted RA, Masi CM, Cacioppo JT. Loneliness predicts increased blood pressure: 5-year cross-lagged analyses in middle-aged and older adults. Psychol Aging. 2010 Mar;25(1):132-41. doi: 10.1037/a0017805. PMID 20230134
- [Background] Hawkley L, Preacher K, Cacioppo J. As We Said, Loneliness (Not Living Alone) Explains Individual Differences in Sleep Quality: Reply. Health Psychol. 2011 Mar;30(2):136. doi: 10.1037/a0022366. No abstract available. PMID 25067871
- [Background] Hobfoll, S. E. (1998). The Plenum series on stress and coping.Stress, culture, and community: The psychology and philosophy of stress. Plenum Press. https://doi.org/10.1007/978-1-4899- 0115-6
- [Background] Holmes EA, O'Connor RC, Perry VH, Tracey I, Wessely S, Arseneault L, Ballard C, Christensen H, Cohen Silver R, Everall I, Ford T, John A, Kabir T, King K, Madan I, Michie S, Przybylski AK, Shafran R, Sweeney A, Worthman CM, Yardley L, Cowan K, Cope C, Hotopf M, Bullmore E. Multidisciplinary research priorities for the COVID-19 pandemic: a call for action for mental health science. Lancet Psychiatry. 2020 Jun;7(6):547-560. doi: 10.1016/S2215-0366(20)30168-1. Epub 2020 Apr 15. PMID 32304649
- [Background] Hulley, S. B., Cummings, S. R., Browner, W. S., Grady, D., Hearst, N., & Newman, T. B. (2007). Designing clinical research. Philadelphia.
- [Background] Insana SP, Hall M, Buysse DJ, Germain A. Validation of the Pittsburgh Sleep Quality Index Addendum for posttraumatic stress disorder (PSQI-A) in U.S. male military veterans. J Trauma Stress. 2013 Apr;26(2):192-200. doi: 10.1002/jts.21793. Epub 2013 Mar 19. PMID 23512653
- [Background] Jansoon, M., & Rello, J. (2020). Mental Health in Healthcare Workers and the Covid-19 Pandemic Era: Novel Challenge for Critical Care Abstract. Journal of Intensive and Critical Care, 6(26), 1-3. https://doi.org/10.36648/2471-8505.6.2.6
- [Background] Lazarus, R. S., & Folkman, S. (1984). Stress, appraisal, and coping. Springer publishing company.
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Kurina LM, Knutson KL, Hawkley LC, Cacioppo JT, Lauderdale DS, Ober C. Loneliness is associated with sleep fragmentation in a communal society. Sleep. 2011 Nov 1;34(11):1519-26. doi: 10.5665/sleep.1390. PMID 22043123
- [Background] Muller AE, Hafstad EV, Himmels JPW, Smedslund G, Flottorp S, Stensland SO, Stroobants S, Van de Velde S, Vist GE. The mental health impact of the covid-19 pandemic on healthcare workers, and interventions to help them: A rapid systematic review. Psychiatry Res. 2020 Nov;293:113441. doi: 10.1016/j.psychres.2020.113441. Epub 2020 Sep 1. PMID 32898840
- [Background] Pfefferbaum B, North CS. Mental Health and the Covid-19 Pandemic. N Engl J Med. 2020 Aug 6;383(6):510-512. doi: 10.1056/NEJMp2008017. Epub 2020 Apr 13. No abstract available. PMID 32283003
- [Background] Poonian J, Walsham N, Kilner T, Bradbury E, Brooks K, West E. Managing healthcare worker well-being in an Australian emergency department during the COVID-19 pandemic. Emerg Med Australas. 2020 Aug;32(4):700-702. doi: 10.1111/1742-6723.13547. Epub 2020 Jun 25. PMID 32386263
- [Background] Rajkumar RP. COVID-19 and mental health: A review of the existing literature. Asian J Psychiatr. 2020 Aug;52:102066. doi: 10.1016/j.ajp.2020.102066. Epub 2020 Apr 10. PMID 32302935
- [Background] Rossi R, Socci V, Pacitti F, Di Lorenzo G, Di Marco A, Siracusano A, Rossi A. Mental Health Outcomes Among Frontline and Second-Line Health Care Workers During the Coronavirus Disease 2019 (COVID-19) Pandemic in Italy. JAMA Netw Open. 2020 May 1;3(5):e2010185. doi: 10.1001/jamanetworkopen.2020.10185. PMID 32463467
- [Background] Shah K, Kamrai D, Mekala H, Mann B, Desai K, Patel RS. Focus on Mental Health During the Coronavirus (COVID-19) Pandemic: Applying Learnings from the Past Outbreaks. Cureus. 2020 Mar 25;12(3):e7405. doi: 10.7759/cureus.7405. PMID 32337131
- [Background] Shaukat N, Ali DM, Razzak J. Physical and mental health impacts of COVID-19 on healthcare workers: a scoping review. Int J Emerg Med. 2020 Jul 20;13(1):40. doi: 10.1186/s12245-020-00299-5. PMID 32689925
- [Background] Shechter A, Diaz F, Moise N, Anstey DE, Ye S, Agarwal S, Birk JL, Brodie D, Cannone DE, Chang B, Claassen J, Cornelius T, Derby L, Dong M, Givens RC, Hochman B, Homma S, Kronish IM, Lee SAJ, Manzano W, Mayer LES, McMurry CL, Moitra V, Pham P, Rabbani L, Rivera RR, Schwartz A, Schwartz JE, Shapiro PA, Shaw K, Sullivan AM, Vose C, Wasson L, Edmondson D, Abdalla M. Psychological distress, coping behaviors, and preferences for support among New York healthcare workers during the COVID-19 pandemic. Gen Hosp Psychiatry. 2020 Sep-Oct;66:1-8. doi: 10.1016/j.genhosppsych.2020.06.007. Epub 2020 Jun 16. PMID 32590254
- [Background] Skinner EA, Zimmer-Gembeck MJ. The development of coping. Annu Rev Psychol. 2007;58:119-44. doi: 10.1146/annurev.psych.58.110405.085705. PMID 16903804
- [Background] Spoorthy MS, Pratapa SK, Mahant S. Mental health problems faced by healthcare workers due to the COVID-19 pandemic-A review. Asian J Psychiatr. 2020 Jun;51:102119. doi: 10.1016/j.ajp.2020.102119. Epub 2020 Apr 22. PMID 32339895
- [Background] Worldometer. (n.d.). Coronavirus Cases. Retrieved August 22, 2020, https://www.worldometers.info /coronavirus/.